CLINICAL TRIAL: NCT03944850
Title: Evaluating the Utility of a Brief Computerized Anxiety Sensitivity Intervention for Opioid Use Disorders: A Pilot Investigation
Brief Title: Computerized Anxiety Sensitivity Treatment for Opioid Use Disorders
Acronym: CAST-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Collaborators: South Central Mental Illness Research, Education & Clinical Center (Unknown)
Responsible Party: Principal Investigator, Amanda M. Raines, Research Psychologist, Southeast Louisiana Veterans Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 365
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Opioid Use Disorder
Keywords: veterans; anxiety sensitivity; opioid use disorder; intervention
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Anxiety Sensitivity Treatment (Experimental): CAST is a newly developed computerized intervention designed to closely model the educational and behavioral techniques that are commonly used in the treatment of anxiety and related conditions.The one time intervention takes approximately 45 minutes to complete.
  Interventions: Behavioral: Computerized Anxiety Sensitivity Treatment

INTERVENTIONS:
Behavioral: Computerized Anxiety Sensitivity Treatment — CAST is a newly developed computerized intervention designed to closely model the educational and behavioral techniques that are commonly used in the treatment of anxiety and related conditions. A psychoeducation component focuses on the nature of anxiety and its effects on the mind and body. Veterans will be taught that physiological and psychological arousal is not dangerous, although they may have developed a conditioned fear of this arousal. Interoceptive exposure (IE) exercises will also be introduced to as a way to reduce or eliminate the conditioned fear response.

SUMMARY:
The primary aim of the current project is to test the acceptability and feasibility of a computerized intervention, titled Computerized Anxiety Sensitivity Treatment (CAST), delivered to Veterans seeking treatment for an opioid use disorder. The second aim of the study is to examine the utility of CAST by gathering data on symptom change. The final aim of the current study is to test the effects of CAST on rates of attendance and retention in a substance use disorder treatment (SUDT) program.

DETAILED DESCRIPTION:
The pilot project will examine the effects of a brief, one-session computerized intervention delivered to Veterans seeking treatment for an opioid use disorder. The opioid epidemic in the United States (US) is having a disproportionate impact on Veterans. Indeed, Veterans are twice as likely to die from an accidental opioid overdose than members of the general population, even after accounting for gender and age distribution. Although many individuals with an opioid addiction seek treatment, a large proportion drop out prematurely and/or relapse, highlighting the need to identify modifiable factors that may contribute to this process. One variable that may be useful in understanding attrition in addiction treatment is anxiety sensitivity (AS). AS is a well-established psychological risk factor reflecting the tendency to fear anxious arousal due to the belief that this arousal will have harmful physical, mental, and/or social consequences. AS is elevated in opioid use populations and predicts treatment dropout among opioid users. Importantly, research suggests that AS is highly malleable. Despite this, to our knowledge no published research to date has systematically explored the utility of AS reduction protocols among opioid users. The first aim of the current project is to test the acceptability and feasibility of a brief, one-session Computerized AS Treatment (CAST) delivered to Veterans seeking treatment for an opioid use disorder. Because this is a pilot project and the study will likely be underpowered to detect treatment effects, we will not emphasize symptom reduction. Nevertheless, a second aim of the current project is to examine the utility of CAST by gathering data on symptom change. Finally, a third aim of the current project is to examine the effects of CAST on rates of attendance and retention in a substance use disorder treatment (SUDT) program.

ELIGIBILITY:
Inclusion Criteria:

* Veterans must be diagnosed with an opioid use disorder

Exclusion Criteria:

* Less than 18 years of age
* Actively suicidal
* Actively psychotic
* Uncontrolled bipolar disorder (i.e., not stable on medications for at least one month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability Questionnaire (IAQ) | One week post-intervention
  The IAQ is an 11-item self-report questionnaire designed to measure treatment satisfaction. The IAQ includes nine items assessing acceptability (e.g., Do you think the information provided during the computerized intervention was helpful? How likely are you to use the information and techniques you learned during the computerized intervention?), which are rated on a 4-point Likert-type scale (0 = no; 1 = somewhat; 2 = moderately; 3 = yes) and two free response items requesting suggestions for improving the treatment. The IAQ will be administered at post-intervention to allow us to assess treatment acceptability.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline
  The AUDIT is a 10-item self-report questionnaire designed by the World Health Organization to classify individuals with alcohol-related problems. The AUDIT will be administered at baseline for descriptive purposes.
Drug Use Disorders Identification Test (DUDIT) | Baseline
  The DUDIT is an 11-item self-report questionnaire intended for use with the AUDIT as a way to classify individuals with drug-related problems. The DUDIT will be administered at baseline for descriptive purposes
PTSD Checklist for DSM-5 (PCL-5) | Baseline
  The PCL-5 is a 20-item self-report questionnaire designed to assess DSM-5 symptoms of PTSD. The PCL-5 will be administered at baseline for descriptive purposes.
Anxiety Sensitivity Index-3 (ASI-3) | Baseline, One week post-intervention, and Four weeks post-intervention
  The ASI-3 is an 18-item self-report questionnaire designed to measure fear of and concern about the negative effects of anxious arousal. The ASI-3 will be administered at all timepoints to allow us to assess treatment-related changes in AS.
Depression Anxiety Stress Scale (DASS) | Baseline, One week post-intervention, and Four weeks post-intervention
  The DASS is a 21-item self-report questionnaire assessing depression, anxiety, and stress symptoms. The DASS will be administered at all timepoints to allow us to assess treatment-related changes in depression, anxiety, and stress symptoms.
Depression Symptom Inventory-Suicide Subscale (DSI-SS) | Baseline, One week post-intervention, and Four weeks post-intervention
  The DSI-SS is a four-item self-report questionnaire designed to assess suicidal ideation, suicidal plans, control of suicidal thoughts, and suicidal impulses. The DSI-SS will be administered at all timepoints to allow us to assess treatment-related changes in suicidality.
Desires for Drug Questionnaire (DDQ) | Baseline, One week post-intervention, and Four weeks post-intervention
  The DDQ is a 13-item self-report questionnaire designed to measure instant (i.e., present moment) cravings associated with opioid use. The DDQ will be administered at all timepoints to allow us to assess treatment-related changes in cravings.
Obsessive Compulsive Drug Use Scale (OCDUS) | Baseline, One week post-intervention, and Four weeks post-intervention
  The OCDUS is a 12-item self-report questionnaire designed to assess heroin thoughts and interference, intention to use heroin and control of its consumption, and resistance against thoughts and decisions to use heroin. The OCDUS will be administered at all timepoints to allow us to assess treatment related changes in thoughts and control over thoughts.
Short Opiate Withdrawal Scale (SOWS) | Baseline, One week post-intervention, and Four weeks post-intervention
  The SOWS is a 10-item self-report questionnaire designed to assess various symptoms of opiate withdrawal. The SOWS will be administered at all timepoints to allow us to assess treatment-related changes in withdrawal symptoms.
Work and Social Adjustment Scale (WSAS) | Baseline, One week post-intervention, and Four weeks post-intervention
  The WSAS is a 5-item descriptive measure of subjective interference of psychiatric symptoms in various life domains (e.g., work, leisure, and family). The WSAS will be administered at all timepoints to allow us to assess treatment-related changes in global life domains.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Raines, PhD, Principal Investigator — Southeast Louisiana Veterans Health Care System
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Data sets underlying this project will not be shared outside the VA, except as required under the Freedom of Information Act (FOIA), for a number of reasons. First, data will be used by the research team to answer additional research questions. Further, veterans may be hesitant to participate in research in which the data will be shared outside the VA and this may act as a barrier to participation and/or benefit from treatment.

REFERENCES:
- [Background] Bohnert AS, Valenstein M, Bair MJ, Ganoczy D, McCarthy JF, Ilgen MA, Blow FC. Association between opioid prescribing patterns and opioid overdose-related deaths. JAMA. 2011 Apr 6;305(13):1315-21. doi: 10.1001/jama.2011.370. PMID 21467284
- [Background] Bohnert AS, Ilgen MA, Galea S, McCarthy JF, Blow FC. Accidental poisoning mortality among patients in the Department of Veterans Affairs Health System. Med Care. 2011 Apr;49(4):393-6. doi: 10.1097/MLR.0b013e318202aa27. PMID 21407033
- [Background] Veilleux JC, Colvin PJ, Anderson J, York C, Heinz AJ. A review of opioid dependence treatment: pharmacological and psychosocial interventions to treat opioid addiction. Clin Psychol Rev. 2010 Mar;30(2):155-66. doi: 10.1016/j.cpr.2009.10.006. Epub 2009 Oct 30. PMID 19926374
- [Background] Reiss, S. and R. McNally, Expectancy model of fear, in Theoretical Issues in Behavior Therapy, S. Reiss and R. Bootzin, Editors. 1985, Academic Press: San Diego, CA. p. 107-122.
- [Background] Lejuez CW, Paulson A, Daughters SB, Bornovalova MA, Zvolensky MJ. The association between heroin use and anxiety sensitivity among inner-city individuals in residential drug use treatment. Behav Res Ther. 2006 May;44(5):667-77. doi: 10.1016/j.brat.2005.04.006. Epub 2005 Jul 5. PMID 16002042
- [Background] Hearon BA, Calkins AW, Halperin DM, McHugh RK, Murray HW, Otto MW. Anxiety sensitivity and illicit sedative use among opiate-dependent women and men. Am J Drug Alcohol Abuse. 2011 Jan;37(1):43-7. doi: 10.3109/00952990.2010.535581. Epub 2010 Nov 19. PMID 21090958
- [Background] Lejuez CW, Zvolensky MJ, Daughters SB, Bornovalova MA, Paulson A, Tull MT, Ettinger K, Otto MW. Anxiety sensitivity: a unique predictor of dropout among inner-city heroin and crack/cocaine users in residential substance use treatment. Behav Res Ther. 2008 Jul;46(7):811-8. doi: 10.1016/j.brat.2008.03.010. Epub 2008 Mar 28. PMID 18466878
- [Background] Schmidt NB, Capron DW, Raines AM, Allan NP. Randomized clinical trial evaluating the efficacy of a brief intervention targeting anxiety sensitivity cognitive concerns. J Consult Clin Psychol. 2014 Dec;82(6):1023-33. doi: 10.1037/a0036651. Epub 2014 May 12. PMID 24821096
- [Background] Schmidt NB, Norr AM, Allan NP, Raines AM, Capron DW. A randomized clinical trial targeting anxiety sensitivity for patients with suicidal ideation. J Consult Clin Psychol. 2017 Jun;85(6):596-610. doi: 10.1037/ccp0000195. Epub 2017 Mar 13. PMID 28287798
- [Background] Barlow, D.H., et al., Behavioral treatment of panic disorder. Behavior Therapy, 1989. 20(2): p. 261-282.
- [Background] Keough ME, Schmidt NB. Refinement of a brief anxiety sensitivity reduction intervention. J Consult Clin Psychol. 2012 Oct;80(5):766-72. doi: 10.1037/a0027961. Epub 2012 Apr 2. PMID 22468909
- [Background] Schmidt NB, Eggleston AM, Woolaway-Bickel K, Fitzpatrick KK, Vasey MW, Richey JA. Anxiety Sensitivity Amelioration Training (ASAT): a longitudinal primary prevention program targeting cognitive vulnerability. J Anxiety Disord. 2007;21(3):302-19. doi: 10.1016/j.janxdis.2006.06.002. Epub 2006 Aug 4. PMID 16889931